CLINICAL TRIAL: NCT07146438
Title: Precision Medicine for OCD - Biobehavioral Tracking of Transcranial Magnetic Stimulation (TMS) With Exposure and Response Prevention (ERP) for Refractory OCD
Brief Title: Transcranial Magnetic Stimulation and Psychotherapy for Treating Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Frank (Other)
Responsible Party: Sponsor-Investigator, Adam Frank, Assistant Professor of Clinical Psychiatry and the Behavioral Sciences, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-24-00659
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: TMS; Transcranial Magnetic Stimulation; OCD; Obsessive Compulsive Disorder; Obsessive-Compulsive Disorder; rTMS; repetitive Transcranial Magnetic Stimulation; psychotherapy; ERP; Magventure; Mental Disorders; Inhibitory Learning; Exposure and Response Prevention
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder; Mental Disorders | interventions — Transcranial Magnetic Stimulation; Palliative Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: All participants will receive repetitive Transcranial Magnetic Stimulation (rTMS). Participants will be randomized to either receive concurrent Exposure and Response Prevention (ERP) Therapy or Supportive Therapy (ST).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will know which treatment group they are in but will be blinded to study hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rTMS+ERP (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Exposure and Response Prevention (ERP) Therapy
- rTMS+ST (Placebo Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Supportive Therapy (ST)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS will be delivered with the MagPro X100 system equipped with a Cool-DB80 coil and a Localite neuronavigation system. Neuronavigation will be performed for anatomical landmarking and co-registration of the brain to Talairach stereotaxic space, with the co-registered coil vertex coordinate (x0, y+60, z+60) as performed in previously published work on dmPFC-rTMS and which represents ~25% of the nasion-inion distance. Posterior coil handle orientation will be used with stimulation parameters of 20Hz repetition rate, 2 second stimulation duration, 20 second inter-train interval, and 50 trains, for a total of 2000 pulses per day. Stimulation will be delivered at 100% of extensor hallucis longus muscle resting motor threshold (MT), as determined by the PI. rTMS will be delivered 5 days per week (Monday through Friday) for 6 weeks for a total of 30 treatment sessions, in keeping with established protocols. Trained research staff will perform daily rTMS treatments and monitor participants.
Behavioral: Supportive Therapy (ST) — Supportive therapy (ST) is a nondirective "talk therapy" focused on enhancing coping skills, strengthening existing resources, and improving daily functioning. Core techniques will include active listening, encouragement, validation, reframing, clarification (summarizing and paraphrasing), and naming problems. Participants will receive two ST sessions per week during the 6-week rTMS course. General goals include using the therapeutic relationship to foster adaptation, improve self-esteem, and support overall well-being. Each session will last 53-60 minutes and take place concurrently with rTMS, with the participant remaining in the TMS treatment room throughout.
  Arms: rTMS+ST
Behavioral: Exposure and Response Prevention (ERP) Therapy — ERP is a form of cognitive-behavioral therapy designed to reduce obsessive-compulsive symptoms by weakening the association between feared stimuli and maladaptive responses. It promotes the formation and recall of non-threatening associations to counter fear-based learning. The participant and therapist will collaboratively create a hierarchy of OCD triggers, rated using the Subjective Units of Distress Scale (SUDS). ERP will begin with exposures rated 4-7 on the SUDS, while participants refrain from engaging in compulsions. Each trigger will be repeated until the SUDS rating decreases by at least 50% before progressing to the next item. Between-session ERP homework will be assigned, and participants will be provided self-monitoring homework rating forms to complete for subsequent review with the therapist. Each ERP session will last 53-60 minutes and will be conducted concurrently with rTMS, with the participant remaining in the TMS treatment room throughout.
  Arms: rTMS+ERP

SUMMARY:
This study will test how people with OCD respond to a type of noninvasive brain stimulation, repetitive Transcranial Magnetic Stimulation (rTMS), when it is combined with psychotherapy. Participants will either engage in Exposure and Response Prevention (ERP) Therapy or supportive therapy (ST) while receiving rTMS. Biobehavioral data from wearable devices and smartphones will be collected to better predict treatment responses. Participants will also undergo repeat resting state functional Magnetic Resonance Imaging (rsfMRI) in order to assess neural predictors and mechanisms of treatment response.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot study to evaluate the feasibility, tolerability, and preliminary effects of combining repetitive transcranial magnetic stimulation (rTMS) with one of two types of therapy for adults with Obsessive-Compulsive Disorder (OCD). All participants will receive rTMS targeted to a specific brain area (the dorsomedial prefrontal cortex/anterior cingulate cortex) five days per week (Monday through Friday) for six weeks, utilizing the FDA-cleared treatment protocol. In addition, participants will receive either Exposure and Response Prevention (ERP), a form of cognitive behavioral therapy, or supportive therapy (ST), delivered virtually twice per week during the rTMS treatment period.

The study lasts a total of 16 weeks. During the first week, participants will complete baseline assessments, including questionnaires about symptoms, functioning, quality of life, and treatment priorities. Participants will undergo a brain scan (rsfMRI) and receive a Fitbit device (Charge 6) to wear throughout the study. Participants will also be guided on how to complete daily self-report check-ins using their smartphone. These check-ins, along with the Fitbit, will collect information about behavior (e.g., sleep, physical activity), physiology (e.g., heart rate), and lived experience (e.g., stress, mood, and symptoms) throughout the study period.

rTMS treatment begins in week 2 and continues for six weeks. ERP or supportive therapy sessions are scheduled twice per week, on the same days as rTMS (Tuesdays and Thursdays), and take place while participants are receiving rTMS in the treatment room. Weekly assessments of OCD symptom severity will be conducted throughout the six-week treatment phase.

After the treatment phase ends in week 8, participants will repeat the brain scan and complete final symptom and functioning assessments. At this time, Fitbit data collection and daily surveys will cease. At week 16 (two months after treatment ends), participants will complete a follow-up assessment to evaluate longer-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obsessive-Compulsive Disorder (OCD) as determined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria.
* Live in Southern California and be willing to attend in-person to receive repetitive Transcranial Magnetic Stimulation (rTMS) 5 times per week for 6 weeks.
* Have completed a prior course of Exposure and Response Prevention (ERP) therapy (at least ten sessions)
* Currently take or have previously tried Serotonin Reuptake Inhibitor (SRI) medication for OCD
* Willing to maintain psychotropic medication levels throughout the 16 weeks of the study

Exclusion Criteria:

* Primary psychiatric diagnosis other than OCD
* Active substance use disorder
* Active suicidality
* Active psychosis
* History of seizures
* Severe neurological impairment
* Pregnant or planning to become pregnant
* Received a prior rTMS course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) Score | From enrollment to end of study at 16 weeks.
  The investigators will use the Yale-Brown Obsessive-Compulsive Scale (YBOCS), the gold standard measure of OCD severity, to assess symptom levels. The YBOCS scale assesses five domains of obsessive and compulsive symptoms, which are each scored on a four-point scale, with 0 being "no symptoms" and 4 being "extreme symptoms". Combined scores range from 0 (no symptoms) to 40 (severe symptoms). A trained clinician, blinded to participant treatment, will administer the YBOCS at study enrollment, weekly during rTMS, at study end, and at 2-month follow-up to determine rate of change of YBOCS score, overall change after treatment, and durability of change at follow-up. Greater decreases in YBOCS scores sustained over time represent a better outcome.

SECONDARY OUTCOMES:
Resting state functional connectivity | From enrollment to the end of treatment at 8 weeks.
  Resting state BOLD-signal fluctuations between hypothesis-driven brain regions-dmPFC (defined as center of mass = MNI X 0, Y+38, Z+24 in MNI-152) and bilateral caudate nucleus (defined as MNI X -8, Y+14, Z+6 and X+6, Y+14, Z+8)-will allow for calculation of functional connectivity between regions. The investigators will calculate change in functional connectivity from baseline to post-treatment.
Recruitment rate | From screening to enrollment.
  Recruitment rate will be calculated as the percentage of individuals enrolled in the study relative to total participants screened.
Adverse and serious adverse event rates | From enrollment to end of study at 16 weeks.
  All adverse and serious adverse events will be recorded for each participant. Differences between treatment groups will be compared.
Study dropout rate | From enrollment to end of study at 16 weeks.
  Rate of dropout from the study will be calculated for all treatment groups as number of individuals starting the study relative to those completing the study. Differences between groups will be compared.
Stanford Expectations of Treatment Scale (SETS) | Assessed at study start; 1 session.
  SETS is a six-item scale used to determine positive and negative perspectives and expectations for treatment before participants begin treatment. Participants are asked to rate how much they agree with a statement based on a seven-point Likert-style scale. Responses are used to assess both positive and negative expectancy for treatment outcomes. The investigators will analyze results overall, based on treatment group, and based on response status.
Self-report priorities in treatment | Assessed at study start; 1 session.
  The investigators will ask participants about their goals for treatment in the current study and their longer-term goals for treatment of OCD. Clinicians will ask about past treatments and provide participants space for free response to be completed via REDCap Survey.
Fidelity of Adherence to Therapy | From start of therapy at week 2 to end of therapy at end of week 7.
  Therapist fidelity, including ratings of therapist adherence and therapist competence to Exposure Response Prevention (ERP) therapy and Supportive Therapy (ST) manuals, and treatment differentiation will be monitored by supervising therapist via video from randomly recorded sessions, stored only until ratings are made. The assessments for the 3 components of treatment fidelity are derived from validated scales and tailored specifically for the elements of ERP and ST included in the treatment manuals for this study (a common practice for clinical research using specific treatment intervention modalities). When deviations from the manualized treatment are noted, supervising therapist will provide feedback and further training to the therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Adam C. Frank, MD, PhD, Principal Investigator — Keck School of Medicine of USC
Locations (1):
- University of Southern California Health Sciences Campus, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No